CLINICAL TRIAL: NCT06327139
Title: A Phase 3 Study Optimising Patient Experience in Head and Neck Radiotherapy
Brief Title: Optimising Patient Experience in Head and Neck Radiotherapy
Acronym: OPEN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Irish Research Radiation Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL 23-24
Record Dates: First submitted 2023-11-20; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Head and Neck Cancer
Keywords: Radiation Therapy; Set-up Accuracy; Faceless Mask; Immobilisation; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a phase III, randomized, single-centre, multiple arm trial of immobilization methods for head and neck cancer patients receiving radical radiation therapy. A faceless three point head and neck mask in conjunction with intra fraction surface guided monitoring, a faceless five point mask in conjunction with intra fraction surface guided monitoring and a conventional closed face five point mask without the use of intra fraction surface guided monitoring are being investigated in this study. The set-up accuracy will be based on the magnitude of the translational corrections measured prior to delivery of each radiation therapy fraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm One: Conventional 5 point closed face immobilisation mask. (Active Comparator): Participants will be immobilized using the standard of care immobilization for patients receiving radical radiation therapy to the head and neck which is a five point closed face mask. The thermoplastic mask immobilizes the patients head, neck and shoulders fully. Participants randomized to this group will not be monitored using intra fraction surface guided monitoring.
  Interventions: Device: Conventional 5 point closed face immobilisation mask.
- Arm Two: 5 point open face immobilization mask (Experimental): Participants will be immobilized using the 5 point open face immobilization mask. The thermoplastic mask immobilizes the participants head, neck and shoulders however the mask does not cover the patients anterior portion of the participants face or chest Participants randomized to this group will be monitored using intra fraction surface guided monitoring.
  Interventions: Device: 5 point open face immobilization mask
- Arm Three: 3 point open face immobilization mask (Experimental): Participants will be immobilized using the 3 point open face immobilization mask. The thermoplastic mask immobilizes the patients head only and does not cover the participants face. Participants randomized to this group will be monitored using intra fraction surface guided monitoring.
  Interventions: Device: 3 point open face immobilization mask

INTERVENTIONS:
Device: Conventional 5 point closed face immobilisation mask. — The conventional closed face mask is a standard of care immobilization device for head and neck cancer patients which covers and immobilizes the entire anterior portion of the patients head, neck and shoulders using a semi rigid thermoplastic material.
  Arms: Arm One: Conventional 5 point closed face immobilisation mask.
Device: 5 point open face immobilization mask — The 5 point open face mask is a type of immobilization device for head and neck cancer patients which does not cover the patients face or chest. The device uses a semi rigid thermoplastic material and covers from the superior aspect of the patients head to the level of their clavicle.
  Other Names: The open face mask is a type of immobilization device for head and neck cancer patients which does not cover the patients face or chest.
  Arms: Arm Two: 5 point open face immobilization mask
Device: 3 point open face immobilization mask — The 3 point open face mask is a type of immobilization device for head and neck cancer patients which does not cover the patients face. The device uses a semi rigid thermoplastic material and covers from the superior aspect of the patients head to the below the patients chin. The three point mask does not cover the patients shoulders and does not extend inferiorly to the level of the clavicle.
  Arms: Arm Three: 3 point open face immobilization mask

SUMMARY:
This study is a phase III, randomized, single-centre, multiple arm trial examining the set-up accuracy of three different types of immobilization methods for head and neck cancer patients receiving radical radiation therapy. The methods of immobilization under investigation in this study are two types of open faced head and neck masks compared with the convention closed faced head and neck mask. Patients receiving treatment using an open faced mask will have their intra fraction motion monitored through the use of intra fraction surface guided monitoring. The study aims to determine the set-up accuracy of the three types of immobilization through measuring the magnitude of the translational corrections on the daily cone beam computed tomography (CBCT). To be eligible for the study a patient must be planned to receive a minimum of 30 fractions of head and neck radiation therapy.

Patients distress levels associated with each type of immobilization device will be measured using the psychological measure General Health Questionnaire-12 (GHQ-12) which will be collected at the beginning and end of their course of radiation therapy treatment.

DETAILED DESCRIPTION:
This study is a phase III, randomized, single-centre, multiple arm trial of immobilization methods for head and neck cancer patients receiving radical radiation therapy.

The two types of immobilization under investigation consist of a faceless three point head and neck mask in conjunction with intra fraction surface guided monitoring and a faceless five point mask in conjunction with intra fraction surface guided monitoring.

The standard of care immobilization consists of a conventional closed face five point mask without the use of intra fraction surface guided monitoring. .

The primary aim of this study is to determine the set-up accuracy of the two types of faceless mask compared with the conventional closed face mask. The set-up accuracy will be measured based on the magnitude of the translational corrections measured prior to delivery of each radiation therapy fraction. This will be measured in millimeters on the daily CBCT.

The secondary aim of this study is to determine the level of distress associated with each type of immobilization device.

A total of 198 evaluable patients will be required for the study. The sample size was calculated based on power calculations to detect clinically significant differences in setup accuracy and patient experience across the three arms.

The enrollment period is expected to be 1 year.

Translational corrections will be measured prior to each fraction of radiation therapy delivered and a minimum of 30 fractions must be delivered in order for a patient to be considered evaluable on trial. The open faced masks will be considered equivalent to the standard of care closed faced mask in terms of set-up accuracy if the difference in translational corrections across the three groups does not indicate a necessity for an increase in the planning target volume for patients planned for radiation therapy treatment using an open faced mask.

Level's of distress will be measured using the psychological measure General Health Questionnaire-12 (GHQ-12). The open faced masks will be considered equivalent to the standard of care closed faced mask the difference in level's of distress between groups does not meet the significance level 0.5.

ELIGIBILITY:
Inclusion Criteria:

1. All radical H&N patients receiving 30-35 fractions of Radiotherapy
2. Written informed consent obtained prior to any study-specific procedures
3. ≥18 years of age

Exclusion Criteria:

1) Patient who from the outset who would not tolerate or would be unable to proceed with treatment if placed in a closed mask, at the discretion of either the patient or the clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The setup accuracy of each immobilization device will be measured based on the magnitude of the translational corrections measured in millimeters prior to delivery of each radiation therapy fraction. | 21 months
  The vertical, lateral and longitudinal translational corrections are measured in millimeters on the daily pre treatment CBCT. The magnitude of this translational correction will be measured for every fraction of radiation therapy and used as a measurement of the set up accuracy of each type of immobilization device under investigation. The mean (M) and standard deviation (SD) of the corrections of the three arms in the translational direction will be analyzed, using Independent t-test and Mann-Whitney U test

SECONDARY OUTCOMES:
Estimate of distress levels during the first week and during the final week of the participants course of radiation therapy using the psychological measure General Health Questionnaire-12 (GHQ-12). | 21 months
  The mean and standard deviation of the GHQ-12 at first week and final week of treatment will be reported. Scoring will be in line with the published guidelines and will use the GHQ-12 summary score. The scales are from 1(Much less than usual) to 4(More so than usual) with 1 being the worst outcome and from 1(Much less able) to 4 (More so than usual) with 1 being the worst outcome. The proportion of patients who report 'More so than usual' for each domain or measure will be reported. Changes in scores over time for each patient will be calculated by subtracting the results at first week of treatment from the last week of treatment results. The mean and SD of the changes will be reported. A Wilcoxon signed rank test will be used to compare differences from baseline. The number of patients who had a clinically meaningful change in distress levels as identified by the method recommended by the EORTC QoL Group at the time of analysis will also be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's Radiation Oncology Network, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No